CLINICAL TRIAL: NCT00612170
Title: A 14-week, Randomized, Double-blind, Placebo-controlled, Multi-center Study of [S,S]-Reboxetine (PNU-165442G) Administered Once Daily (O.D.) in Patients With Fibromyalgia
Brief Title: A 14-week, Multi-center Study of [S,S]-Reboxetine in Patients With Fibromyalgia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6061043; A6061043
Record Dates: First submitted 2008-01-29; First posted 2008-02-11 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Fibromyalgia
Keywords: Phase 3, safety and efficacy study, [S,S[-Reboxetine, Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — O-methyl reboxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 3 (Experimental)
  Interventions: Drug: [S,S]-Reboxetine
- 4 (Sham Comparator)
  Interventions: Drug: Placebo
- 1 (Experimental)
  Interventions: Drug: [S,S]-Reboxetine
- 2 (Experimental)
  Interventions: Drug: [S,S]-Reboxetine

INTERVENTIONS:
Drug: [S,S]-Reboxetine — 10 mg oral tablet once a day dosing
  Arms: 3
Drug: Placebo — 0 mg oral tablet once a day dosing
  Arms: 4
Drug: [S,S]-Reboxetine — 4 mg oral tablet once a day dosing
  Arms: 1
Drug: [S,S]-Reboxetine — 8 mg oral tablet once a day dosing
  Arms: 2

SUMMARY:
This is a study to investigate the effectiveness and safety of [S,S]-Reboxetine in relieving the symptoms of Fibromyalgia in patients. A previous study demonstrated clinically meaningful treatment effects in fibromyalgia, based on pain and functional endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of any race, at least 18 years of age
* Patients must meet the ACR criteria for fibromyalgia (ie, widespread pain present for at least 3 months, and pain in at least 11 of 18 specific tender point sites)

Exclusion Criteria:

* Patients with other severe pain (eg, Diabetic Peripheral Neuropathy and PostHerpetic Neuralgia) that may confound assessment or self evaluation of the pain associated with fibromyalgia
* Patients with any autoimmune rheumatic disorder, non-focal rheumatic disease (other than fibromyalgia), active infection, or untreated endocrine disorder
* A current or recent diagnosis (last 6 months) or episode of major depressive disorder, dysthymia and/or uncontrolled depression
* History of mania, hypomania, other psychotic disorder, or current mood disorder with psychotic features

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1129 (Actual)
Dates: Start 2007-12; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the endpoint mean pain score | 14 weeks
Fibromyalgia Impact Questionnaire | 14 weeks

SECONDARY OUTCOMES:
Change from baseline in the endpoint mean sleep interference score | 14 weeks
Patient Global Impression of Change | 14 weeks
Multidimensional Assessment of Fatigue | 14 weeks
Hospital Anxiety and Depression Scale | 14 weeks
Short Form 36 | 14 weeks
Sheehan Disability Score | 14 weeks
Pain Visual Analogue Scale | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (122):
- United States (114):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Huntsville, Alabama
  - Pfizer Investigational Site, Tallassee, Alabama
  - Pfizer Investigational Site, Chandler, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Carmichael, California
  - Pfizer Investigational Site, Elk Grove, California
  - Pfizer Investigational Site, Fullerton, California
  - Pfizer Investigational Site, Lafayette, California
  - Pfizer Investigational Site, Northridge, California
  - Pfizer Investigational Site, Oceanside, California
  - Pfizer Investigational Site, Roseville, California
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, San Jose, California
  - Pfizer Investigational Site, Santa Ana, California
  - Pfizer Investigational Site, New London, Connecticut
  - Pfizer Investigational Site, Brooksville, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Sarasota, Florida
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, Sunrise, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Venice, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Winter Haven, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Aurora, Illinois
  - Pfizer Investigational Site, Gurnee, Illinois
  - Pfizer Investigational Site, Moline, Illinois
  - Pfizer Investigational Site, Oak Brook, Illinois
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Dubuque, Iowa
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Pratt, Kansas
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Madisonville, Kentucky
  - Pfizer Investigational Site, Mount Sterling, Kentucky
  - Pfizer Investigational Site, Baton Rouge, Louisiana
  - Pfizer Investigational Site, Wheaton, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Brockton, Massachusetts
  - Pfizer Investigational Site, Fall River, Massachusetts
  - Pfizer Investigational Site, North Dartmouth, Massachusetts
  - Pfizer Investigational Site, Watertown, Massachusetts
  - Pfizer Investigational Site, Wellesley Hills, Massachusetts
  - Pfizer Investigational Site, Worcester, Massachusetts
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Chaska, Minnesota
  - Pfizer Investigational Site, Edina, Minnesota
  - Pfizer Investigational Site, Rochester, Minnesota
  - Pfizer Investigational Site, Olive Branch, Mississippi
  - Pfizer Investigational Site, Columbia, Missouri
  - Pfizer Investigational Site, Jefferson City, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Henderson, Nevada
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Brooklyn, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, The Bronx, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Salisbury, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, Toledo, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Bend, Oregon
  - Pfizer Investigational Site, Eugene, Oregon
  - Pfizer Investigational Site, Medford, Oregon
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Altoona, Pennsylvania
  - Pfizer Investigational Site, Bethlehem, Pennsylvania
  - Pfizer Investigational Site, Bridgeville, Pennsylvania
  - Pfizer Investigational Site, Duncansville, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, West Reading, Pennsylvania
  - Pfizer Investigational Site, Willow Grove, Pennsylvania
  - Pfizer Investigational Site, Cumberland, Rhode Island
  - Pfizer Investigational Site, Lincoln, Rhode Island
  - Pfizer Investigational Site, Warwick, Rhode Island
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Bristol, Tennessee
  - Pfizer Investigational Site, Jackson, Tennessee
  - Pfizer Investigational Site, Johnson City, Tennessee
  - Pfizer Investigational Site, Kingsport, Tennessee
  - Pfizer Investigational Site, Milan, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Beaumont, Texas
  - Pfizer Investigational Site, Bryan, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, DeSoto, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Lake Jackson, Texas
  - Pfizer Investigational Site, Nassau Bay, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Ogden, Utah
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Arlington, Virginia
  - Pfizer Investigational Site, Charlottesville, Virginia
  - Pfizer Investigational Site, Virginia Beach, Virginia
  - Pfizer Investigational Site, Kirkland, Washington
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Spokane, Washington
  - Pfizer Investigational Site, Milwaukee, Wisconsin
  - Pfizer Investigational Site, Oregon, Wisconsin
- Canada (8):
  - Pfizer Investigational Site, Kelowna, British Columbia
  - Pfizer Investigational Site, Bathurst, New Brunswick
  - Pfizer Investigational Site, Moncton, New Brunswick
  - Pfizer Investigational Site, Hawkesbury, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Pointe-Claire, Quebec
  - Pfizer Investigational Site, Québec, Quebec
  - Pfizer Investigational Site, Sherbrooke, Quebec

REFERENCES:
- [Derived] Arnold LM, Hirsch I, Sanders P, Ellis A, Hughes B. Safety and efficacy of esreboxetine in patients with fibromyalgia: a fourteen-week, randomized, double-blind, placebo-controlled, multicenter clinical trial. Arthritis Rheum. 2012 Jul;64(7):2387-97. doi: 10.1002/art.34390. PMID 22275142
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6061043&StudyName=A%2014-week%2C%20multi-center%20study%20of%20%5BS%2CS%5D-Reboxetine%20in%20patients%20with%20Fibromyalgia.